CLINICAL TRIAL: NCT05070676
Title: Accuracy of a Newly Developed Mobile Application Versus the Conventional Method of Cephalometric Analysis in the Diagnosis of Dental and Skeletal Deformities Among Pre-adolescent Patients: A Diagnostic Accuracy Study
Brief Title: Accuracy of a Newly Developed Mobile Application Versus the Conventional Method of Cephalometric Analysis in the Diagnosis of Dental and Skeletal Deformities Among Pre-adolescent Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nehal Mohamed Mostafa Ahmed, principal investigator, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: mobile app in ceph.analysis
Record Dates: First submitted 2021-09-14; First posted 2021-10-07 (Actual); Last update posted 2021-10-07 (Actual); Status verified 2021-09

CONDITIONS: Mobile Application; Cephalometric Analysis

STUDY DESIGN:
Intervention Model Description: A newly developed mobile application will be developed to help pedodontists in orthodontic diagnosis, and treatment of dentoalveolar, or skeletal deformations
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lateral cephalometric radiographs of pre-adolescent patients (8-13) years old. (Experimental)
  Interventions: Diagnostic Test: newly developed mobile application

INTERVENTIONS:
Diagnostic Test: newly developed mobile application — The application will be developed in native Android, using Java (backend) and XML (front-end) as the programming language. The program of choice will be Android Studio®, YouTube® (video reproduction) and Firebase® (database) will be used as external APIs (Application Programming Interfaces).
  The layout of the application will be developed using:
  Adobe Illustrator® software. The logo, brand, objects, and shapes of the mobile application will be designed to enable to resize of the images without any loss of quality, due to the wide range of scales available in current smartphones

SUMMARY:
This study aims to evaluate the accuracy of a newly developed mobile application versus the conventional method of cephalometric analysis in the diagnosis of dental and skeletal deformities among pre-adolescent patients.

DETAILED DESCRIPTION:
A mobile application will be developed to help pedodontists in orthodontic diagnosis, and treatment of dentoalveolar, or skeletal deformations ,The mobile application will provide quick cephalometric analysis and therefore, offers rapid and accurate case diagnosis, reduces errors in tracing, measurement, and identification of the landmark.

Reference test: Cephalometric analysis by the conventional method

-Trial design: Diagnostic accuracy study

ELIGIBILITY:
Inclusion Criteria:

1. Digital Lateral cephalometric radiographs of pre-adolescent patients (8-13) years old.
2. Cephalogram of good quality with all landmarks clearly visible
3. Presence of central incisors and first molars on cephalogram
4. Cephalogram with teeth in maximum intercuspation

Exclusion Criteria:

-

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 17 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2022-11-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
The Accuracy of the newly developed mobile application versus the conventional method of cephalometric analysis in the diagnosis | 3 monthes
  The accuracy of the mobile application will be measured based on cephalometric analysis angles( by degrees) of Egyptian people according to Soliman SA. PHD thesis 1988